CLINICAL TRIAL: NCT00548132
Title: Reducing Catheter-Related Bloodstream Infections in the ICU With a Chlorhexidine-Impregnated Sponge (BIOPATCH)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00424-0805-01 (BJH Foundation); WUSM HRPO# 05-1186
Record Dates: First submitted 2007-10-22; First posted 2007-10-23 (Estimated); Results first posted 2013-08-22 (Estimated); Last update posted 2013-09-12 (Estimated); Status verified 2013-08

CONDITIONS: Catheter-related Bloodstream Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (No Intervention): Patients in this arm will continue to get routine care
- Chlorhexidine-impregnated foam dressing (Experimental): Patient's catheters were cleaned with chlorhexidine-alcohol solution at least weekly before application of the Biopatch. These were evaluated daily and if the dressing was bloody, soiled or damaged, the dressing and the Biopatch were replaced prior to the 7-day period.
  Interventions: Device: Chlorhexidine-impregnated foam dressing

INTERVENTIONS:
Device: Chlorhexidine-impregnated foam dressing — Patients in the treatment arm will have the Biopatch incorporated into their catheter care protocol. ICU nurses were instructed on the proper use of this novel dressing/sponge. Catheter dressing changes will only be done every 7 days unless there is visible blood, soiling underneath the dressing, or if the dressing comes off.
  Other Names: Biopatch Antimicrobial Dressing
  Arms: Chlorhexidine-impregnated foam dressing

SUMMARY:
We proposed to perform a prospective randomized controlled trial to study the effect of the use of a commercially-available chlorhexidine-impregnated sponge (Biopatch) as part of central venous catheter care on catheter-related bloodstream infections among patients in two Barnes-Jewish Hospital ICUs.

DETAILED DESCRIPTION:
At the time of the inception of this study, there were no published randomized controlled trial on the efficacy of the Biopatch in reducing bloodstream infections. Preliminary data has shown that the Biopatch decreases colonization of the catheter exit site and thereby decrease bloodstream infections but this was at that time only theoretical.

ELIGIBILITY:
Inclusion Criteria:

* patients who are admitted to the ICU with a central venous catheter (i.e. triple lumen catheters, quadruple lumen catheters, percutaneously inserted central catheters, arterial catheters, intraaortic balloon pumps, Swan-Ganz catheters).

Exclusion Criteria:

* patients who are not enrolled into the trial within 7 days of having the catheter being placed and patients who are allergic to chlorhexidine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1088 (Actual)
Dates: Start 2006-02; Primary Completion 2008-02 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bernard C Camins, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Barnes- Jewish Hospital, St Louis, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The patients were recruited from two ICUs at BJH. The nurse was asked to page the research coordinators on patients who were scheduled to have a central venous catheter placed for IV access.
Pre-assignment Details: Patients or family member authorized to consent for the patient (if the patient was not competent to consent to the study) were approached by study personnel for inclusion into the study. Written informed consent was obtained for all subjects and randomization group was assigned in blocks of 4.
Groups:
- Standard of Care: Patients in this arm will continue to get the standard catheter care protocol without the use of the chlorhexidine-impregnated foam dressing.
Period: Overall Study
Arm/Group | Standard of Care | Chlorhexidine-impregnated Foam Dressing
Started | 534 | 554
Consented to Study | 534 | 554
Completed | 534 | 554
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Chlorhexidine-impregnated Foam Dressing: Patients in this group had the Biopatch applied on the catheter exit site after insertion of the catheter. Dressings were changed every 7 days along with the Biopatch after the skin was cleaned with a chlorhexidine-alcohol antiseptic solution. Dressings were assessed daily and changed if they were soiled, non-intact, or bloody before the 7-day period was up.
- Total: Total of all reporting groups
Arm/Group | Standard of Care | Chlorhexidine-impregnated Foam Dressing | Total
Number analyzed (Participants) | 534 | 554 | 1088
Age Continuous [Mean (Standard Deviation); unit: years] — Age at enrollment was collected for this measure
  years | 58.26 (16.88) | 58.70 (16.83) | 58.47 (16.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 304 | 325 | 629
  Male | 230 | 229 | 459
Region of Enrollment [Number; unit: participants]
  United States | 534 | 554 | 1088

OUTCOME MEASURES:

1. Primary Outcome: The Number of Catheter Related Bloodstream Infections (BSI) /1000 Catheter Days in Both Arms
Description: The outcome measure is the number of episodes of bloodstream infections (BSI) divided by the catheter days at risk multiplied by 1000 for standardization
Time Frame: 2 years
Population: Based on previous data (unpublished),there would be a 60% reduction in the incidence of bloodstream infections-- the primary outcome. The number of patients included in this study had a large enough sample size to show a statistical difference.
Measure: Number; unit: BSIs /1000 catheter days
Groups:
- Standard of Care: Standard of care
- Chlorhexidine Impregnated Sponge: Patients in this group had the Biopatch applied on the catheter exit site after insertion of the catheter. Dressings were changed every 7 days along with the Biopatch after the skin was cleaned with a chlorhexidine-alcohol antiseptic solution. Dressings were assessed daily and changed if they were soiled, non-intact, or bloody before the 7-day period was up.
Arm/Group | Standard of Care | Chlorhexidine Impregnated Sponge
Number analyzed (Participants) | 534 | 554
BSIs /1000 catheter days | 4.74 | 4.72
Statistical Analysis 1: Comparison: Standard of Care vs Chlorhexidine Impregnated Sponge; The null hypothesis is that the Bloostream infection per 1000 catheter days will be similar in both groups. In 2004, 6122 catheter days occurred in by both ICUs. If 15% of these were excluded, then 5203 catheter days/year will be eligible for analysis. The difference in infection rates will reach statistical significance at 12 months with a P-value of 0.04. At 24 months, the P-value will be more significant at 0.006; Test type: Superiority or Other; p = 0.05, Cochran-Mantel-Haenszel; This was calculated based on the assumption that only 85% of eligible patients will consent to the study; Risk Ratio (RR) = 0.46, 95% CI 2-sided [0.24 to 0.90], Standard Deviation 0.05 — The standard of care is the numerator and the intervention group is the denominator

2. Secondary Outcome: Clinical Sepsis Episodes/Per 1000 Catheter Days
Description: This measure is a combination of patients with positive blood cultures (BSI) and patients who had signs and symptoms of sepsis but with negative blood cultures. These patients still required treatment with antibiotics.
Time Frame: 2 years
Measure: Number; unit: sepsis episodes/1000 catheter days
Groups:
- Standard of Care: Standard catheter care-use of chlorhexidine-alcohol solution to prep the catheter site and then a bioocclusive dressing is applied
- Intervention Group: Patients in this group had the Biopatch applied on the catheter exit site after insertion of the catheter. Dressings were changed every 7 days along with the Biopatch after the skin was cleaned with a chlorhexidine-alcohol antiseptic solution. Dressings were assessed daily and changed if they were soiled, non-intact, or bloody before the 7-day period was up.
Arm/Group | Standard of Care | Intervention Group
Number analyzed (Participants) | 534 | 554
sepsis episodes/1000 catheter days | 7.8 | 8.5

ADVERSE EVENTS:
Arm/Group | Standard of Care | Chlorhexidine-impregnated Foam Dressing
Serious Adverse Events (participants affected / at risk) | 0/534 | 0/554
Other Adverse Events (participants affected / at risk) | 0/534 | 0/554

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No